CLINICAL TRIAL: NCT01877304
Title: Effect of Drug Targeting Nebulization on Lung Deposition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AKITA
Record Dates: First submitted 2013-05-29; First posted 2013-06-13 (Estimated); Last update posted 2013-06-13 (Estimated); Status verified 2013-06

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AKITA with program central deposition (Experimental): Nebulization for central deposition
  Interventions: Device: AKITA
- AKITA with program for peripheral deposition (Active Comparator): Nebulization for peripheral deposition
  Interventions: Device: AKITA

INTERVENTIONS:
Device: AKITA

SUMMARY:
To compare deposition between two modalities of nebulization

ELIGIBILITY:
Inclusion Criteria:

* Free of respiratory disease

Exclusion Criteria:

* Smokers

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2010-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Lung deposition by scintigraphy | After 15 minutes

SECONDARY OUTCOMES:
Regional deposition by scintigraphy | After 15 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium